CLINICAL TRIAL: NCT03241342
Title: Double-Blind, Placebo-Controlled, Parallel Design, Phase 2 Study to Assess Clinical Activity and Safety of Enobosarm (GTx-024) in Postmenopausal Women With Stress Urinary Incontinence
Brief Title: Study to Assess Enobosarm (GTx-024) in Postmenopausal Women With Stress Urinary Incontinence
Acronym: ASTRID
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GTx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: G201002
Record Dates: First submitted 2017-08-02; First posted 2017-08-07 (Actual); Results first posted 2020-11-12 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — ostarine

STUDY DESIGN:
Intervention Model Description: Double-blind, placebo-controlled, parallel design, randomized, multicenter, Phase 2 study consisting of the following periods: screening period, treatment period, and follow-up period.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 1 mg GTx-024 (Active Comparator): Study drug will be provided as softgel capsules in blister packaging, labeled and designed to protect study blinding. All subjects will take 2 softgel capsules orally, once daily.
  Interventions: Drug: GTx 024
- 3 mg GTx-024 (Active Comparator): Study drug will be provided as softgel capsules in blister packaging, labeled and designed to protect study blinding. All subjects will take 2 softgel capsules orally, once daily.
  Interventions: Drug: GTx 024
- matching placebo (Placebo Comparator): Study drug will be provided as softgel capsules in blister packaging, labeled and designed to protect study blinding. All subjects will take 2 softgel capsules orally, once daily.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GTx 024 — Study drug is an opaque, white to off-white, size 5, oval Softgel capsule containing the active ingredient GTx-024.
  Other Names: Enobosarm
  Arms: 1 mg GTx-024; 3 mg GTx-024
Drug: Placebo — Placebo study drug is identical in appearance to the GTx-024 study drug and contains polyethylene glycol 400 but not GTx-024.
  Arms: matching placebo

SUMMARY:
GTx-024 is an orally bioavailable and tissue-selective nonsteroidal selective androgen receptor modulator (SARM) that has demonstrated androgenic and anabolic activity and is currently being evaluated as a potential treatment for stress urinary incontinence (SUI) in postmenopausal women. Urinary incontinence and pelvic floor disorders are major health problems for women, especially as they age. Pelvic floor muscle relaxation has been found to correlate with lower urinary tract symptoms including SUI. Muscles of the pelvic floor and lower urinary tract are crucial for supporting the pelvic organs and micturition; however, damage to the muscles or lack of hormonal stimulation are thought to contribute to pelvic organ prolapse and urinary incontinence. Although anabolic steroids may increase muscle mass and strength, lack of oral bioavailability and known potential risks have limited their use. Nonsteroidal SARMs have potential to achieve benefits of anabolic steroid therapy (improved muscle mass, cholesterol/triglyceride levels, glucose metabolism, and bone density) with fewer adverse effects, such as hirsutism and acne, in women. Both nonclinical and clinical data suggest that SARMs may provide a new therapeutic option for pelvic floor and lower urinary tract disorders, as both testosterone and its more potent metabolite, dihydrotestosterone, have anabolic effects on muscle.

ELIGIBILITY:
Key Inclusion Criteria:

* SUI symptoms of at least 6 months duration
* Predominant SUI as determined at the Screening Visit using the Medical, Epidemiological, and Social Aspects of Aging (MESA) urinary questionnaire.
* 24-Hour pad weight > 3 g during the screening period
* A minimum of 1 and no more than 15 SUI episodes on any single day AND no fewer than 9 total SUI episodes over 3 days during the screening period
* Positive bladder stress test conducted during the Screening Visit

Key Exclusion Criteria:

* History of pelvic radiation treatment
* History of urethral diverticula
* History of urethral sling or anterior prolapse repair
* Treatment with urethral bulking agents and/or other SUI procedure or surgery within the 6 months prior to the Screening Visit
* Known vesicoureteral reflux, vaginal prolapse beyond the introitus, or other significant pelvic floor abnormalities
* Urinary incontinence of neurogenic etiology
* Morbidly obese (defined as 100 pounds over ideal body weight, or body mass index 40 or greater)
* Chronic hepatitis
* Hepatic cirrhosis
* Evidence of active infection with hepatitis B or hepatitis C
* History of human immunodeficiency virus (HIV) infection
* Subjects with a history of breast or endometrial cancer

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female, 18 to 80 years of age, inclusive, at screening; having undergone spontaneous, medically induced, or surgical menopause prior to the start of the study
Enrollment: 491 (Actual)
Dates: Start 2017-08-21 (Actual); Primary Completion 2018-09-21 (Actual); Study Completion 2018-09-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth M Peters, MD, Principal Investigator — Oakland University, William Beaumont School of Medicine
Locations (62):
- United States (62):
  - Urology Center of Alabama, Homewood, Alabama
  - Coastal Clinical Research Inc, Mobile, Alabama
  - Alaska Clinical Research Center, Anchorage, Alaska
  - Mayo Clinic Arizona, Phoenix, Arizona
  - Urological Associates of Southern Arizona, Tucson, Arizona
  - Women's Healthcare Research Corporation, San Diego, California
  - American Institute of Research, Whittier, California
  - Genitourinary Surgical Consultants, Denver, Colorado
  - Urology Associates Research, Englewood, Colorado
  - Women's Health Specialty Care, Farmington, Connecticut
  - Coastal Connecticut Research, LLC, New London, Connecticut
  - Bladder Control Center of Connecticut, Norwalk, Connecticut
  - James A Simon MD PC, Washington D.C., District of Columbia
  - South Florida Medical Research, Aventura, Florida
  - Tampa Bay Medical Research Inc, Clearwater, Florida
  - Midland Florida Clinical Research Center LLC, DeLand, Florida
  - Precision Clinical Research, Lauderdale Lakes, Florida
  - Lone Star Research Center, Miami, Florida
  - Medical Research of Florida, Miami, Florida
  - Clinical Research Center of Florida, Pompano Beach, Florida
  - Mount Vernon Clinical Research LLC, Sandy Springs, Georgia
  - Clinical Research Prime, Idaho Falls, Idaho
  - Idaho Urologic Institue, Meridian, Idaho
  - Women's Health Institution of Illinois, Oak Lawn, Illinois
  - First Urology PSC, Jeffersonville, Indiana
  - Iowa Clinic, West Des Moines, Iowa
  - DelRicht Clinical Research, LLC, New Orleans, Louisiana
  - Regional Urology, Shreveport, Louisiana
  - Chesapeake Urology Associates PA, Hanover, Maryland
  - Boston Clinical Trials, Boston, Massachusetts
  - Bay State clinical Trials, Watertown, Massachusetts
  - Beyer Research, Kalamazoo, Michigan
  - William Beaumont Hospital Urology Research, Royal Oak, Michigan
  - Women's Clinic of Lincoln, Lincoln, Nebraska
  - Sheldon J Freedman MD Ltd, Las Vegas, Nevada
  - Premier Urology Group, LL, Edison, New Jersey
  - Lawrence Obs Gyn clinical Research, Lawrenceville, New Jersey
  - Delaware Valley Urology, Mount Laurel, New Jersey
  - Accumed Research Associates, Garden City, New York
  - Manhattan Medical Research Practice PLLC, New York, New York
  - Premier Medical Group, Poughkeepsie, New York
  - Circuit Clinical, West Seneca, New York
  - American Health Research Inc, Charlotte, North Carolina
  - Alliance Urology Specialist PA, Greensboro, North Carolina
  - Eastern Carolina Women's, New Bern, North Carolina
  - The Urology Group, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Aventiv Research, Columbus, Ohio
  - Institute for Female Pelvic Medicine, Allentown, Pennsylvania
  - Urologic Consultants of Southeastern PA LLP, Bala-Cynwyd, Pennsylvania
  - University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - Carolina Urologic Research, Myrtle Beach, South Carolina
  - The Jackson Clinic, Jackson, Tennessee
  - Elligo - Austin Area OBGYN, Austin, Texas
  - Urology Clinics of North Texas, Dallas, Texas
  - Clinical Trials of Texas Incorporated, San Antonio, Texas
  - Urology San Antonio Research PA, San Antonio, Texas
  - Synexus Clinical Research Advantage, Inc. - Wasatch Peak Family Practice, Layton, Utah
  - Urology of Virginia, Virginia Beach, Virginia
  - Urology Northwest PS, Mountlake Terrace, Washington
  - Seattle Womens: Health, Research, Gynocology, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 1 mg GTx-024 | 3 mg GTx-024 | Matching Placebo
Started | 163 | 163 | 165
Completed | 141 | 132 | 138
Not Completed | 22 | 31 | 27
Not completed — Adverse Event | 5 | 8 | 4
Not completed — Lack of Efficacy | 0 | 0 | 1
Not completed — noncompliance with study drug | 2 | 1 | 1
Not completed — sponsor decision | 0 | 1 | 2
Not completed — not reported | 15 | 21 | 19

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 mg GTx-024 | 3 mg GTx-024 | Matching Placebo | Total
Number analyzed (Participants) | 163 | 163 | 165 | 491
Age, Continuous [Median (Full Range); unit: years] | 60 [42 to 80] | 59 [40 to 79] | 58 [44 to 80] | 59 [40 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 163 | 163 | 165 | 491
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 10 | 15 | 38
  Not Hispanic or Latino | 149 | 152 | 150 | 451
  Unknown or Not Reported | 1 | 1 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 2 | 1 | 6
  Asian | 1 | 1 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 25 | 20 | 12 | 57
  White | 131 | 139 | 150 | 420
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 1 | 0 | 4
Baseline number of stress incontinence episodes per day [Mean (Full Range); unit: episodes per day] | 4.588 [3 to 11.67] | 4.329 [3 to 12.67] | 4.459 [3 to 12] | 4.4 [3 to 12.67]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a ≥ 50% Reduction From Baseline in the Mean Number of Stress Incontinence Episodes Per Day at Week 12
Description: Mean number of subject-reported stress incontinence episodes per day through a responder analysis, where a responder is defined as having a ≥ 50% reduction at the end of treatment (Week 12) compared to baseline in the number of stress incontinence episodes
Time Frame: 12 Weeks
Population: full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | 1 mg GTx-024 | 3 mg GTx-024 | Matching Placebo
Number analyzed (Participants) | 163 | 163 | 165
Participants | 94 | 96 | 87

ADVERSE EVENTS:
Time Frame: 7 months
Arm/Group | 1 mg GTx-024 | 3 mg GTx-024 | Matching Placebo
All-Cause Mortality (participants affected / at risk) | 0/163 | 0/163 | 0/165
Serious Adverse Events (participants affected / at risk) | 3/163 | 2/163 | 4/165
Other Adverse Events (participants affected / at risk) | 105/163 | 104/163 | 96/165
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 1 mg GTx-024 (N=163) | 3 mg GTx-024 (N=163) | Matching Placebo (N=165)
acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0
goiter (Endocrine disorders) | 0 | 1 | 0
abscessed limb (Infections and infestations) | 0 | 0 | 1
osteomyelitis (Infections and infestations) | 0 | 0 | 1
hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
spinal disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
cerebral vascular accident (Nervous system disorders) | 0 | 1 | 0
pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
dysaesthesia (Nervous system disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 1 mg GTx-024 (N=163) | 3 mg GTx-024 (N=163) | Matching Placebo (N=165)
anemia (Blood and lymphatic system disorders) | 0 | 1 | 0
lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1
polycythaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
thrombocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0
acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0
cardiomegaly (Cardiac disorders) | 1 | 0 | 0
palpitations (Cardiac disorders) | 1 | 1 | 0
ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 1
motion sickness (Ear and labyrinth disorders) | 0 | 0 | 1
vertigo (Ear and labyrinth disorders) | 1 | 0 | 0
goiter (Endocrine disorders) | 0 | 1 | 0
hypothyroidism (Endocrine disorders) | 1 | 0 | 0
blepharitis (Eye disorders) | 1 | 1 | 0
chalazion (Eye disorders) | 1 | 0 | 0
dry eye (Eye disorders) | 0 | 0 | 1
eye discharge (Eye disorders) | 0 | 1 | 0
eye pain (Eye disorders) | 1 | 0 | 0
eye swelling (Eye disorders) | 1 | 0 | 0
vision blurred (Eye disorders) | 2 | 0 | 1
visual impairment (Eye disorders) | 0 | 0 | 1
abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1
abdominal distension (Gastrointestinal disorders) | 2 | 0 | 2
abdominal hernia (Gastrointestinal disorders) | 1 | 0 | 0
abdominal pain (Gastrointestinal disorders) | 2 | 1 | 2
abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 2
abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1
change of bowel habit (Gastrointestinal disorders) | 0 | 0 | 1
colitis (Gastrointestinal disorders) | 0 | 0 | 1
constipation (Gastrointestinal disorders) | 4 | 3 | 3
diarrhea (Gastrointestinal disorders) | 2 | 3 | 5
diverticulum (Gastrointestinal disorders) | 1 | 0 | 0
dry mouth (Gastrointestinal disorders) | 1 | 5 | 4
dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1
eructation (Gastrointestinal disorders) | 1 | 0 | 0
flatulence (Gastrointestinal disorders) | 1 | 0 | 2
food poisoning (Gastrointestinal disorders) | 1 | 0 | 0
gastritis (Gastrointestinal disorders) | 1 | 0 | 1
hemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0
nausea (Gastrointestinal disorders) | 4 | 4 | 7
oesophageal stenosis (Gastrointestinal disorders) | 1 | 0 | 0
vomiting (Gastrointestinal disorders) | 2 | 0 | 1
chest pain (General disorders) | 1 | 0 | 0
cyst (General disorders) | 0 | 1 | 0
energy increased (General disorders) | 0 | 0 | 1
fatigue (General disorders) | 2 | 3 | 3
feeling abnormal (General disorders) | 0 | 0 | 1
feeling hot (General disorders) | 0 | 1 | 1
hypothermia (General disorders) | 0 | 1 | 0
influenza like illness (General disorders) | 1 | 1 | 0
malaise (General disorders) | 1 | 0 | 0
non cardiac chest pain (General disorders) | 1 | 0 | 0
oedema peripheral (General disorders) | 7 | 3 | 1
peripheral swelling (General disorders) | 1 | 1 | 0
polyp (General disorders) | 0 | 1 | 0
pyrexia (General disorders) | 1 | 0 | 0
thirst (General disorders) | 0 | 0 | 1
hypersensitivity (Immune system disorders) | 0 | 0 | 1
abscess limb (Infections and infestations) | 0 | 0 | 1
acute sinusitis (Infections and infestations) | 1 | 0 | 0
bronchitis (Infections and infestations) | 3 | 3 | 3
candida infection (Infections and infestations) | 0 | 1 | 0
cellulitis (Infections and infestations) | 1 | 0 | 1
clostridium difficile infection (Infections and infestations) | 0 | 0 | 1
diverticulitis (Infections and infestations) | 1 | 0 | 0
ear infection (Infections and infestations) | 1 | 0 | 0
escherichia (Infections and infestations) | 1 | 0 | 1
eye infection (Infections and infestations) | 0 | 0 | 1
fungal infection (Infections and infestations) | 1 | 1 | 0
gastroenteritis (Infections and infestations) | 0 | 2 | 1
gastroenteritis viral (Infections and infestations) | 0 | 0 | 2
genital herpes (Infections and infestations) | 0 | 3 | 0
herpes zoster (Infections and infestations) | 3 | 0 | 0
influenza (Infections and infestations) | 3 | 3 | 3
localized infection (Infections and infestations) | 1 | 0 | 0
mycoplasma infection (Infections and infestations) | 0 | 1 | 0
nasopharyngitis (Infections and infestations) | 4 | 7 | 6
osteomyelitis (Infections and infestations) | 0 | 0 | 1
otitis media acute (Infections and infestations) | 0 | 1 | 0
pharyngitis (Infections and infestations) | 0 | 0 | 1
pneumonia (Infections and infestations) | 1 | 1 | 3
post procedural infection (Infections and infestations) | 0 | 1 | 0
respiratory tract infection viral (Infections and infestations) | 1 | 0 | 0
rhinitis (Infections and infestations) | 0 | 1 | 0
sinusitis (Infections and infestations) | 0 | 2 | 0
streptococcal infection (Infections and infestations) | 0 | 1 | 0
tooth infection (Infections and infestations) | 1 | 1 | 1
upper respiratory tract infection (Infections and infestations) | 7 | 7 | 10
urinary tract infection (Infections and infestations) | 17 | 29 | 18
urinary tract infection fungal (Infections and infestations) | 0 | 1 | 0
vaginal infection (Infections and infestations) | 1 | 1 | 0
viral infection (Infections and infestations) | 0 | 0 | 1
vulvovaginal mycotic infection (Infections and infestations) | 2 | 0 | 1
arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 1
contusion (Injury, poisoning and procedural complications) | 1 | 0 | 1
fall (Injury, poisoning and procedural complications) | 1 | 0 | 1
foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
joint injury (Injury, poisoning and procedural complications) | 0 | 1 | 1
laceration (Injury, poisoning and procedural complications) | 1 | 0 | 1
ligament rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1
ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0
post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0
procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0
radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
soft tissue injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
sternal fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1
tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
alanine aminotransferase increasae (Investigations) | 1 | 1 | 0
aspartate aminotransferase increase (Investigations) | 1 | 1 | 0
blood alkaline phosphatase increase (Investigations) | 1 | 0 | 0
blood creatinine phophokinase mb increase (Investigations) | 1 | 0 | 0
blood creatinine phosphokinase increase (Investigations) | 1 | 0 | 0
blood creatinine decrease (Investigations) | 1 | 0 | 0
blood creatinine increase (Investigations) | 7 | 0 | 1
blood glucose increase (Investigations) | 2 | 0 | 1
blood pressure increase (Investigations) | 0 | 1 | 2
blood urine present (Investigations) | 1 | 0 | 0
c reactive protein increase (Investigations) | 1 | 1 | 0
arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 3 | 3
back pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 2
fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
limb discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 3 | 4
muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
myalgia (Musculoskeletal and connective tissue disorders) | 3 | 1 | 1
neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 3 | 1
poly arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
spinal disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
laryngeal papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
burning sensation (Nervous system disorders) | 0 | 0 | 1
cerebrovascular accident (Nervous system disorders) | 0 | 1 | 1
dizziness (Nervous system disorders) | 4 | 1 | 2
dysaesthesia (Nervous system disorders) | 1 | 0 | 0
dysarthria (Nervous system disorders) | 0 | 0 | 1
headache (Nervous system disorders) | 3 | 12 | 7
memory impairment (Nervous system disorders) | 0 | 1 | 0
migraine (Nervous system disorders) | 1 | 0 | 0
neuropathy peripheral (Nervous system disorders) | 1 | 0 | 0
paraesthesia (Nervous system disorders) | 1 | 0 | 1
sciatica (Nervous system disorders) | 1 | 0 | 0
somnolence (Nervous system disorders) | 1 | 1 | 0
tension headache (Nervous system disorders) | 1 | 0 | 1
affect lability (Psychiatric disorders) | 0 | 1 | 0
agitation (Psychiatric disorders) | 0 | 0 | 2
anger (Psychiatric disorders) | 1 | 0 | 0
anxiety (Psychiatric disorders) | 0 | 1 | 0
attention deficit hyperactivity disorder (Psychiatric disorders) | 1 | 0 | 0
bruxism (Psychiatric disorders) | 0 | 0 | 1
confusional state (Psychiatric disorders) | 0 | 0 | 1
depression (Psychiatric disorders) | 1 | 1 | 0
emotional disorder (Psychiatric disorders) | 0 | 0 | 1
insomnia (Psychiatric disorders) | 0 | 5 | 1
irritability (Psychiatric disorders) | 0 | 1 | 1
libido increase (Psychiatric disorders) | 0 | 1 | 0
mental disorder (Psychiatric disorders) | 0 | 0 | 1
sleep disorder (Psychiatric disorders) | 0 | 0 | 1
azotemia (Renal and urinary disorders) | 1 | 0 | 0
bladder disorder (Renal and urinary disorders) | 1 | 0 | 0
bladder pain (Renal and urinary disorders) | 0 | 1 | 0
contracted bladder (Renal and urinary disorders) | 0 | 0 | 1
dysuria (Renal and urinary disorders) | 1 | 0 | 0
hematuria (Renal and urinary disorders) | 3 | 2 | 3
leukocyturia (Renal and urinary disorders) | 1 | 0 | 0
micturition urgency (Renal and urinary disorders) | 0 | 1 | 0
nephrolithiasis (Renal and urinary disorders) | 2 | 1 | 0
nocturia (Renal and urinary disorders) | 0 | 0 | 1
polyuria (Renal and urinary disorders) | 1 | 0 | 0
stress urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0
urethral caruncle (Renal and urinary disorders) | 0 | 1 | 0
urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0
urinary retention (Renal and urinary disorders) | 1 | 0 | 0
urine odor abnormal (Renal and urinary disorders) | 1 | 0 | 0
breast cyst (Reproductive system and breast disorders) | 0 | 1 | 0
breast tenderness (Reproductive system and breast disorders) | 2 | 2 | 0
clitoral engorgement (Reproductive system and breast disorders) | 0 | 1 | 0
coital bleeding (Reproductive system and breast disorders) | 0 | 0 | 1
cystocele (Reproductive system and breast disorders) | 0 | 1 | 0
endometrial thickening (Reproductive system and breast disorders) | 2 | 1 | 3
hydrometra (Reproductive system and breast disorders) | 3 | 1 | 0
ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 1
pelvic congestion (Reproductive system and breast disorders) | 1 | 0 | 0
pelvic pain (Reproductive system and breast disorders) | 1 | 1 | 2
uterine polyp (Reproductive system and breast disorders) | 1 | 0 | 1
vaginal discharge (Reproductive system and breast disorders) | 2 | 1 | 0
vaginal enlargement (Reproductive system and breast disorders) | 1 | 0 | 0
vaginal hemorrhage (Reproductive system and breast disorders) | 1 | 1 | 1
vaginal lesion (Reproductive system and breast disorders) | 0 | 0 | 1
vulva cyst (Reproductive system and breast disorders) | 0 | 0 | 1
vulvovaginal discomfort (Reproductive system and breast disorders) | 1 | 0 | 0
vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 0 | 1
asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 2
dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0
oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
reflux laryngitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
sleep apnea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
upper airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
acne (Skin and subcutaneous tissue disorders) | 1 | 3 | 3
alopecia (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
hirsutism (Skin and subcutaneous tissue disorders) | 0 | 1 | 3
hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 2
photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 1
rash papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
rosacea (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
seborrhoea (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
skin irritation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
urticaria (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
aortic aneurysm (Vascular disorders) | 0 | 0 | 1
flushing (Vascular disorders) | 0 | 1 | 0
hot flush (Vascular disorders) | 1 | 4 | 0
hypertension (Vascular disorders) | 3 | 6 | 2
hypertensive crisis (Vascular disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (1018-04-10): https://cdn.clinicaltrials.gov/large-docs/42/NCT03241342/Prot_SAP_000.pdf